CLINICAL TRIAL: NCT04157062
Title: An Open-Label Trial of Repetitive Transcranial Magnetic Stimulation for Opioid Use Disorder
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Research never commenced.
Sponsor: West Virginia University (Other)
Responsible Party: Principal Investigator, James Mahoney, Assistant Professor/Clinical Neuropsychologist, West Virginia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1907653805
Record Dates: First submitted 2019-11-06; First posted 2019-11-08 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-03

CONDITIONS: Opioid-use Disorder; Substance-Related Disorders; Chemically-Induced Disorders; Mental Disorder
Keywords: Transcranial Magnetic Stimulation
MeSH Terms: conditions — Opioid-Related Disorders; Substance-Related Disorders; Chemically-Induced Disorders; Mental Disorders | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: This is an open-label study for participants who have opioid use disorder (OUD) that are eligible to have repetitive transcranial magnetic stimulation (rTMS) targeting the left dorsolateral prefrontal cortex (DLPFC).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Study Group (Experimental): Participants will receive a type of TMS called repetitive TMS (rTMS) wherein the magnetic pulses delivered will be close together in a rapid sequence. They will receive excitatory rTMS with a stimulation frequency of 10 Hz or higher.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS)

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation (rTMS) — During the rTMS session, an electromagnetic coil is placed against the subjects scalp. The electromagnet painlessly delivers a magnetic pulse that stimulates nerve cells in the region of the brain involved in memory and thinking.

SUMMARY:
The purpose of this study is to understand the role of repetitive Transcranial Magnetic Stimulation (rTMS) in reducing opioid and other substance use and craving and improving thinking skills.

DETAILED DESCRIPTION:
The overarching goal of this study is to investigate a form of neuromodulation, rTMS, as an adjunctive treatment for OUD by evaluating the impact of rTMS on substance use, craving and inhibitory control, factors which contribute to relapse. The primary outcome will be the assessment of whether rTMS reduces substance use. Additional exploratory outcomes include the assessment of whether rTMS applied to the DLPFC provides neuromodulatory effects through the assessment of craving, inhibitory control, and functional connectivity via MRI. The targeted sample size for this open-label study, where all enrolled subjects will receive 9 sessions of active rTMS over 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide written informed consent, and to comply with study procedures.
* Be actively enrolled in the COAT Program
* Meet DSM-V criteria for a primary OUD assessed via structured clinical interview
* Columbia-Suicide Severity Rating Scale score < 4
* Be abstinent from opioids (other than prescribed buprenorphine/naloxone) and illicit substances other than marijuana at the time of the enrollment, confirmed via urine drug screen
* Willing to practice contraception to avoid pregnancy the duration of the study

Exclusion Criteria:

* Medical conditions that preclude rTMS: including vasodepressor syncope, glaucoma, increased intracranial pressure, cardiac disease, migraine disorder, cerebral vascular events (cerebral vascular accident, transient ischemic attack), any brain lesions (such multiple sclerosis), brain injury, seizure disorder (or family history) of any type, and have cardiac pacemakers or implanted medication pumps
* DSM-V criteria for major psychiatric illness other than depression
* Major Cognitive Disorder (as evidenced by a score of <21/30 on the Mini Mental Status Exam (MMSE)
* Pregnancy
* Positive responses to the TMS Adult Safety Screen or the MRI checklist
* Intracranial metallic objects (excluding dental fillings)
* Uncorrected visual acuity problems
* Mobility limitations
* Clinically significant EKG abnormalities (including QTc interval prolongation >450 ms in men or >480 ms in women)
* Unwillingness to abstain from prescribed drugs
* Prior rTMS treatment
* Other mental or physical conditions that, in the PI's opinion, would be inappropriate for study participation.
* Intake of one or a combination of the following drugs forms a 'Strong Potential Hazard' for application of rTMS due to their significant seizure threshold lowering potential:

  * Imipramine, Amitriptyline, Doxepine, Nortriptyline, Maprotiline, Chlorpromazine, Clozapine, Foscarnet, Ganciclovir, Ritonavir, Amphetamines, Cocaine (MDMA, ecstasy), Phencyclidine (PCP, angel's dust), Ketamine, Gamma-hydroxybutyrate (GHB), Alcohol, Theophylline.
  * The inclusion of a patient on any of the above medication will be carefully evaluated and a decision documented by the medically responsible physician. The risk is dependent on the patient's past medical history, drug dose, speed of dose increase (or decrease), history of recent medication changes or duration of treatment, and combination with other CNS active drugs.
* Recent withdrawal from one of the following drugs forms a 'Strong Relative Hazard' for application of rTMS due to the resulting significant seizure threshold lowering potential:

  * Alcohol, Barbiturates, Benzodiazepines, Meprobamate, Chloral hydrate

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2021-09-30 (Estimated); Primary Completion 2025-03-19 (Actual); Study Completion 2025-03-19 (Actual)

PRIMARY OUTCOMES:
rTMS reduces substance use | 1 - 7 weeks
  Opioid use as measured by quantitative urine toxicology via high pressure liquid chromatography at screening, baseline, enrollment (3 times per week for 3 weeks), and follow-up phases (weekly for 4 weeks).

SECONDARY OUTCOMES:
rTMS applied to the DLPFC provides neuromodulatory effects | 1 - 7 weeks
  Participants will complete standardized measures of mood, drug craving, and executive function at screening, baseline, enrollment (3 times per week for 3 weeks), and follow-up phases (weekly for 4 weeks).

OTHER OUTCOMES:
Functional connectivity changes | week 1, week 3, and week 7
  Measure by MRI scans prior to and following the first rTMS session, following the final rTMS session, and during the final follow-up.